CLINICAL TRIAL: NCT06663410
Title: Sphenopalatine Ganglion Block with Tx360 Nasal Applicator for Trigeminal Neuralgia: a Prospective Observational Study
Brief Title: Sphenopalatine Ganglion Block with Tx360 for Trigeminal Neuralgia
Status: Completed | Type: Observational
Sponsor: Aretaieio Hospital (Other)
Responsible Party: Principal Investigator, Christina Orfanou, Resident anesthesiologist, MD, MSc, Aretaieio Hospital
Other Study IDs: 274/12-11-2020; Aretaieio Hospital (Other: Aretaieio Hospital, NKUA, Greece)
Record Dates: First submitted 2024-10-24; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Trigeminal Neuralgia
Keywords: Trigeminal Neuralgia; SPG block; Tx360; nasal applicator
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Fifteen patients of both sexes, older than 18 years, ASA I or II, TN of any etiology: Patients will undergo bilateral sphenopalatine ganglion block with Tx360 nasal applicator using 0.3cc lidocaine 2% in each side, once every week, for a 6-week period.
  Interventions: Device: SPG block with the use of the Tx360 device

INTERVENTIONS:
Device: SPG block with the use of the Tx360 device — A SPG block was performed using the Tx360 nasal applicator according to the manufacturer's instructions bilaterally, injecting 0.3cc of lidocaine 2% into each nostril.

SUMMARY:
The aim of this study was to investigate the effect of sphenopalatine ganglion (SPG) block bilaterally through a nasal device called Tx360 by delivering 0.3cc of lidocaine 2% for pain relief in patients with Trigeminal Neuralgia (TN).

DETAILED DESCRIPTION:
Trigeminal neuralgia (TN) is a chronic condition that causes sudden, intense facial pain that has a severe impact on patients' life quality and everyday functioning. Even with many treatments available, some patients still struggle to manage their pain effectively.

Sphenopalatine ganglion (SPG) block, delivered through a recently introduced nasal applicator called Tx360, has shown promising results for those patients suffering persistent facial pain, icluding cases of TN.

The purpose of this study was to observe how effective the SPG block delivering lidocaine 2% via the Tx360 is for pain relief in patients with TN. The patients' diagnosis included classical or atypical TN affecting the V2 (maxillary) or V3 (mandibular) branches, with partial or complete resistance to medication.

Researchers measured pain levels using the Numerical Rating Scale (NRS) and evaluated the effects of treatment on patients' physical and mental wellbeing using the Short Form-36 (SF-36) Quality of Life Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* older than 18 years
* ASA I or II
* trigeminal neuralgia of any etiology

Exclusion Criteria:

* anatomical abnormalities of the nasal septum,
* rhinitis or nasal inflammation due to medication,
* nasal septum perforation,
* nasal or paranasal sinus surgery (within the last 3 months)
* dryness or irritation of the nasal mucosa, localized pain, nasal discharge, or bleeding from the nose,
* disorders related to bleeding or coagulation,
* significant respiratory distress,
* presence of malignancies, including angiofibroma or other tumors of the paranasal sinuses, or granulomas,
* persistent nasal congestion lasting more than 10 days, accompanied by high fever, discolored nasal mucosa, or facial pain and headaches,
* nasal or skull fractures occurring within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of both sexes, ASA I or II, with classical or atypical, V2 (maxillary branch) or V3 (mandibular branch) trigeminal neuralgia, partly or completely drug-resistant, with NRS = 8-9, under pharmaceutical treatment, with minimal or no clinical improvement and/or poor patient satisfaction. A written informed consent was obtained from each eligible patient.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
NRS pain score | From enrollment to the end of the follow-up period, which included an initial 6-week period, where the treatment was being administered, and a subsequent 12-week period post-treatment that served for follow-up purposes.
  Outcome measures were assessed on a weekly basis for the initial 6-week treatment period, that is at every visit where SPG block would be administered, and on a monthly basis for the subsequent 12-week follow-up period, where patients participated in scheduled monthly follow-up calls.
  Patients were instructed to maintain a detailed pain diary for these 18 weeks and were asked about their pain intensity as measured with the Numerical Rating Scale (NRS) scoring system.
  NRS consists of a simple 11-point scale from zero to ten, where zero corresponds to non-existent pain and ten corresponds to the worst possible pain the patient has ever experienced. Patients choose the number that best corresponds to the intensity of their pain.

SECONDARY OUTCOMES:
changes in the 9 components measured by the SF-36 questionnaire | during the first visit to the clinic and 3 months after the completion of the treatment
  The SF-36 Quality of Life Questionnaire consists of 36 closed-ended questions, with 2-5 ratings in the answers. Each question contributes to a total score ranging from 0 to 100, measuring both mental and physical health status. This questionnaire is appropriate for self-completion as well as for completion during a telephone or a face-to-face interview, provided that the participant is over 14 years old.
  During the patients' first clinic appointment, they were asked to complete the SF-36 Questionnaire to assess the impact of trigeminal neuralgia on their daily functioning. Three months after the treatment was completed, we conducted a follow-up assessment using the same questionnaire in order to evaluate any changes in the nine components of the SF-36 questionnaire: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, general health, and perceived health change.

CONTACTS AND LOCATIONS:
Overall Officials: Athanasia Tsaroucha, Assoc. Prof., Study Director — Aretaieio Hospital, National and Kapodistrian University of Athens
Locations (1):
- Aretaieio Hospital, National and Kapodistrian University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cady R, Saper J, Dexter K, Manley HR. A double-blind, placebo-controlled study of repetitive transnasal sphenopalatine ganglion blockade with tx360((R)) as acute treatment for chronic migraine. Headache. 2015 Jan;55(1):101-16. doi: 10.1111/head.12458. Epub 2014 Oct 23. PMID 25338927
- [Background] Candido KD, Massey ST, Sauer R, Darabad RR, Knezevic NN. A novel revision to the classical transnasal topical sphenopalatine ganglion block for the treatment of headache and facial pain. Pain Physician. 2013 Nov-Dec;16(6):E769-78. PMID 24284858
- [Background] Ho KWD, Przkora R, Kumar S. Sphenopalatine ganglion: block, radiofrequency ablation and neurostimulation - a systematic review. J Headache Pain. 2017 Dec 28;18(1):118. doi: 10.1186/s10194-017-0826-y. PMID 29285576
- [Background] Piagkou M, Demesticha T, Troupis T, Vlasis K, Skandalakis P, Makri A, Mazarakis A, Lappas D, Piagkos G, Johnson EO. The pterygopalatine ganglion and its role in various pain syndromes: from anatomy to clinical practice. Pain Pract. 2012 Jun;12(5):399-412. doi: 10.1111/j.1533-2500.2011.00507.x. Epub 2011 Sep 29. PMID 21956040